CLINICAL TRIAL: NCT06202495
Title: Dentine Hypersensitivity Treated With Diode Laser and Amino Fluoride: A Randomized Clinical Trial
Brief Title: Dentine Hypersensitivity Treated With Laser and Fluoride.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Professor, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-FLUORIDELASER
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sensitive Dentin
Keywords: Dentine hypersensitivity; fluoride; laser
MeSH Terms: conditions — Dentin Sensitivity | interventions — Lasers; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser and Fluoride (Experimental): The treatment group will be treated with amino-fluoride gel (Elmex Dental Gel, Colgate-Palmolive company, New York, 300 Park Ave, United States) in association 980nm diode laser (doctor smile wiser by Lambda s.p.a. Via dell'Impresa, 1, 36040 Brendola VI, Italy) 1.5 W, pulsed mode 2 mm from tooth surface. For treatment will be used 400 μm diameter and 5 mm long tips of for 4 minutes
  Interventions: Device: Laser and Fluoride
- Fluoride (Active Comparator): The control group will be treated with amino-fluoride gel (Elmex Dental Gel, Colgate-Palmolive company, New York, 300 Park Ave, United States) for 4 minutes.
  Interventions: Other: Fluoride

INTERVENTIONS:
Device: Laser and Fluoride — topic application of amino-fluoride gel (Elmex Dental Gel, Colgate-Palmolive company, New York, 300 Park Ave, United States) in association 980nm diode laser (doctor smile wiser by Lambda s.p.a. Via dell'Impresa, 1, 36040 Brendola VI, Italy) 1.5 W, pulsed mode 2 mm from tooth surface
  Arms: Laser and Fluoride
Other: Fluoride — topic application of amino-fluoride gel (Elmex Dental Gel, Colgate-Palmolive company, New York, 300 Park Ave, United States)
  Arms: Fluoride

SUMMARY:
The aim of the present report is to evaluate the amino fluoride gel with or without application of diode laser on pain due to dentine hypersensitivity.

NRS (numerical rating scale) index will be used to evaluate the pain suffered by each patient after cold air blow stimulus.

After treatment application, the follow-up timing planned for each patient will be at 1 week, 1 month, 3 months and 6 months

DETAILED DESCRIPTION:
The aim of the present report is to evaluate the amino fluoride gel with or without application of diode laser on pain due to dentine hypersensitivity.

The study is designed with a split mouth design. NRS (numerical rating scale) index will be used to evaluate the pain suffered by each patient. The pain response will be stimulated by thermal urge (cold air blow). Teeth will be divided in two groups. The treatment group, treated with 980nm diode laser and amino fluoride gel; the control group, treated only with amino fluoride gel.

The follow-up timing planned for each patient will be at 1 week, 1 month, 3 months and 6 months. In these follow-up sessions a revaluation of the pain response is performed using the NRS index.

ELIGIBILITY:
Inclusion Criteria:

* Teeth in good periodontal health
* Good oral hygiene
* Dentine hypersensitivity: NRS (Numerical Rating Scale) ≥ 3

Exclusion Criteria:

* Teeth local disease or fractures in treatment area
* Irreversible teeth necrosis or pulpitis
* Definitive restorations or veneers
* Recent use of painkillers or anti-inflammatory drugs,
* Treatment for dentine Hypersensitivity less than 6 months before the study start
* Therapies contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
NRS (numerical rating scale) | Before treatment and 1 week, 1 month, 3 months, 6 months after treatment
  The dentine hypersensitivity will be evaluated with the Numerical Rating Scale ( NRS ), where 0 meant pain absence and 10 a unbearable pain (Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, et al. Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011;41(6):1073-93.)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS PhD MSc, Principal Investigator — Unit of Dental Hygiene - Section of Dentistry - Dep of Clin Surg Diagn Ped Sci - University of Pavia
Locations (1):
- A.O. Mater Domini, U.O. Odontoiatria, University of Catanzaro "Magna Græcia"., Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No